CLINICAL TRIAL: NCT04860609
Title: Compare the Effect of Spinal Decompression in Lumber Spine Disc Protrusion Patients
Brief Title: Compare the Effects of Decompression on Lumber Disc Protrusion Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aqua Medical Services (Pvt) Ltd (Industry)
Responsible Party: Principal Investigator, Mir Arif Hussain, Mir Arif Hussain, Aqua Medical Services (Pvt) Ltd
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Abdul Ghaffor 00501
Record Dates: First submitted 2021-04-21; First posted 2021-04-27 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Lumbar Disc Herniation
Keywords: Decompression; Disc herniation; ODI; LBP
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: control group will recevie conventional physiotherapy sessions while the experimental group receive conventional along with decompression
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy (Active Comparator): It includes the pre-physiotherapy session by conventional physiotherapy
  Interventions: Other: Conventional Physiotherapy
- Lumber spinal decompression (Experimental): It includes the pre-physiotherapy session iby lumber spinal decompression along with conventional therapy.
  Interventions: Other: Lumber Spinal Decompression

INTERVENTIONS:
Other: Conventional Physiotherapy — The treatment will be given in the following way.
  1. Tens
  2. Infrared/Moist Heat heat for 10 minutes at low back region.
  3. Lumbar Mobilization (Maitland) CPA 3 sets of 10 reps
  4. Stretching Exercises (Calf, Hams, Back Extensors) 3 sets of 8-10 reps
  5. Strengthening Exercises (Back Extensors) 3 sets of 8-10 reps
  6. Postural Education
  7. Home Plan
  8. Bed Rest with lumbar Sacral Support
  9. Home plan:
  Exercises Posture Correction Precautions Contra indication
  Arms: Conventional Physiotherapy
Other: Lumber Spinal Decompression — The treatment will be given in the following way.
  1. Tens
  2. Infrared/Moist Heat heat for 10 minutes at low back region.
  3. Lumbar Mobilization (Maitland) CPA 3 sets of 10 reps
  4. Stretching Exercises (Calf, Hams, Back Extensors) 3 sets of 8-10 reps
  5. Strengthening Exercises (Back Extensors) 3 sets of 8-10 reps
  6. Postural Education
  7. Home Plan
  8. Decompression therapy session lumbar spinal decompression therapy for 30 minutes.
  9. Home plan:
  Exercises Posture Correction Precautions Contra indication
  Arms: Lumber spinal decompression

SUMMARY:
This is an RCT study in which 60 participant are included and half of the participant are randomized via lottery method in control and experimental group after fulfilling the inclusion criteria. The sampling technique is convenient sampling . The study compare the effects of conventional Physical Therapy and Decompression Therapy and determine the effectiveness of Decompression as treatment procedure for patients with Lumbar disc protrusion. The data collection procedure included the NPRS, ODI, structural questionnaire and assesment on the 1st, 4th and 8th visit. Data will be analyzed on IBM SPSS-21 {Statistical Procedure of Social Sciences} software. The assessment will be done on 1st, 4th and 8th visits. after checking the normality of the date the Parametric/Non Parametric test will be apply to compare the means of the these groups. The 95% confidence interval will be used in term OD p value 0.05

DETAILED DESCRIPTION:
Low back pain is the common problem of our society, 80% people experience back pain at some stage of their life. Low Back pain life time prevalence is 65% to 80% and It is estimated that 28% experience disabling low back pain sometime during their lives.Point prevalence ranged from 12% to 33%, 1-year prevalence ranged from 22% to 65%, and lifetime prevalence ranged from 11% to 84%.Back pain peak prevalence age is 40-50, First episode of start in the 20's and recurrence rates between 39-71%. Women tend to be affected more in cervical spine problem then men and Men tend to more affected in lumbar spine problem than women. Majority (80-90%) of low back disorders occur at the L4/5 and/or L5/S1. The occupational risk factor include driving (P<0.001), lifting, carrying, pulling, pushing, and twisting (P<0.001 for all variables) as well as nondriving vibrational exposure (P<0.001).

Maitland divides lumber spine problems into two groups, in first group the L4/5 and L5/S1 intervertebral discs are frequently a source of symptoms and second group have postural, muscles balance, muscles weakness, muscles spasm degenerative changes and mechanical movement disorders problems. The L5-S1 Segment is the most common site of problem in the spine because this level bears more weight, Center of gravity passes directly through this vertebra, transition L5 Mobile and S1 Stable, Large angle B/w L5 & S1 and great amount of movement.

The intervertebral disk makes up 1/3 of the total length of vertebral column. The disc contains 85% to 90% of water, but the amount decrease up to 65% with age. The water binding capacity of the disc decrease with age and degenerative changes begin to occur after 2nd decade of the life. The Facet joint carry 20-25% axial body load but this may reach 70% with degeneration of the Disc. The most significant biochemical change to occur in disc degeneration is loss of proteoglycan. This loss is responsible for a fall in the osmotic pressure of the disc matrix and therefore a loss of hydration. Loading may thus lead to inappropriate stress concentrations along the endplate or in the annulus.

Decompression therapy is a result oriented approach but it expensive and minimum availability in Pakistan. In physical therapy we use different exercise to solve the multiple spine problems. Some exercise used to treat orthopedic component such as mobilization, manipulation, SNAGS, and traction. Some exercise used to treat myogenic component such as Muscle energy technique, neuromuscular reeducation, active isolated stretch etc. Some exercise used to treat neurogenic component such as Neurodynamics, Active release technique etc. As we know the fascia is important component in our body most of the time the fascia restriction make the patient condition verse. Guy Voyer introduce the systems of exercise more the 35 years ago which works specially on spine at every intervertebral level including costal and pelvic articulation. These exercises are called Elongation Longitudinaux avec Decoaption Osteo-Articulaire (ELDOA) or simply Longitudinal Osteo-Articular De-coaptation Stretching (LOADS). It can be describe as fascial stretch that's localizes tension at the level of a specific spinal segment and create decompression. In which he combined improving the tone of the intrinsic muscles of the spine along with reinforcing the extrinsic muscles related to the spine aim the back and stretching the interlinking paraspinal muscles. ELDOA exercise is design for every level of the spine from base of the skull to sacro iliac joint. In each ELDOA exercise we create fascial tension above and below the joint or disc that one is trying to "open up" or decompress. The outcomes include; Release vertebral compression, improved blood circulation, Disc re-hydration, improve muscle tone and awareness. One of my study also proved that ELDOA Exercises improve the pain and functional level in the spinal disc protrusion patients.

ELIGIBILITY:
Inclusion Criteria:

1. MRI of lumbar spine showing lumbar disc bulge
2. Localized and radiating pain more than 5 on NPRS

Exclusion Criteria

1. Lumbar spondylolisthesis
2. Spinal stenosis
3. Fracture of lumbar spine
4. Spinal tumor
5. Ankylosing spondylitis
6. Patients taking blood thinner medication

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale for back | 8th weeks
  It is numeric pain rating scale for measuring pain intensity. it ranges from 0-10.In which 0 shows no pain,1-3 (mild pain),4-6(moderate pain) and 10 shows severe pain. As guided by the researcher, pain intensity was marked by the patient
Flexion Range of Motion of lumber | 8th weeks
  Double inclinometer is used
SLR | 8th weeks
  Single Inclinometer
Side bending Lumber ROm | 8th week
  Double inclinometer
Extension Lumber ROM | 8th week
  Double inclinometer is used

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghaffor Sajjad, PhD, Principal Investigator — Shifa tameer-e-millat university Islamabad
Locations (1):
- Abdul Ghaffor Sajjad, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] rchaeos Projects. (1999). Preliminary Site Report of the Oriental Institute of the University of Vienna and Archaeos: Excavation Project at Tell Arbid, Sector D Retrieved 04/09/2004, 2004, from http://www.archaeos.org/html/repor2js.htm
- [Background] Atlas SJ, Keller RB, Wu YA, Deyo RA, Singer DE. Long-term outcomes of surgical and nonsurgical management of sciatica secondary to a lumbar disc herniation: 10 year results from the maine lumbar spine study. Spine (Phila Pa 1976). 2005 Apr 15;30(8):927-35. doi: 10.1097/01.brs.0000158954.68522.2a. PMID 15834338
- [Background] Breslau, A. M., & Gabe, M. (1962). Ergebnisse der Polysaccharidhistochemie, Microorganismen, Invertebraten : mit 25. Stuttgart: Fischer.
- [Background] Delauche-Cavallier MC, Budet C, Laredo JD, Debie B, Wybier M, Dorfmann H, Ballner I. Lumbar disc herniation. Computed tomography scan changes after conservative treatment of nerve root compression. Spine (Phila Pa 1976). 1992 Aug;17(8):927-33. PMID 1387974
- [Background] Dvorak J, Valach L, Fuhrimann P, Heim E. The outcome of surgery for lumbar disc herniation. II. A 4-17 years' follow-up with emphasis on psychosocial aspects. Spine (Phila Pa 1976). 1988 Dec;13(12):1423-7. doi: 10.1097/00007632-198812000-00016. PMID 2975065
- [Background] Frymoyer JW, Pope MH, Costanza MC, Rosen JC, Goggin JE, Wilder DG. Epidemiologic studies of low-back pain. Spine (Phila Pa 1976). 1980 Sep-Oct;5(5):419-23. doi: 10.1097/00007632-198009000-00005. PMID 6450452
- [Background] Hammer, W. I. (2007). Functional soft-tissue examination and treatment by manual methods: Jones & Bartlett Learning.
- [Background] Khan, A. G. S. G. A., & Khan, A. (2016). Fascia Stretching Improve the Pain and Functional Level in Disc Protrusion Patients. Journal of Riphah College of Rehabilitaion Sciences, 4(1), 7-10.
- [Background] Krause M, Refshauge KM, Dessen M, Boland R. Lumbar spine traction: evaluation of effects and recommended application for treatment. Man Ther. 2000 May;5(2):72-81. doi: 10.1054/math.2000.0235. PMID 10903582
- [Background] Magee, D. J. (2014). Orthopedic physical assessment: Elsevier Health Sciences. Maitland, G. D., Hengeveld, E., Banks, K., & English, K. (2005). Maitland's vertebral manipulation (Vol. 1): Butterworth-Heinemann.
- [Background] Manchikanti L. Epidemiology of low back pain. Pain Physician. 2000 Apr;3(2):167-92. PMID 16906196
- [Background] Robin, M., & Stephen, M. The lumbar spine mechanical diagnosis & therapy, volume one and two. 2004: Spinal Publications, Nya Zeeland
- [Background] van der Windt DA, Simons E, Riphagen II, Ammendolia C, Verhagen AP, Laslett M, Deville W, Deyo RA, Bouter LM, de Vet HC, Aertgeerts B. Physical examination for lumbar radiculopathy due to disc herniation in patients with low-back pain. Cochrane Database Syst Rev. 2010 Feb 17;(2):CD007431. doi: 10.1002/14651858.CD007431.pub2. PMID 20166095
- [Background] Weber H. Lumbar disc herniation. A controlled, prospective study with ten years of observation. Spine (Phila Pa 1976). 1983 Mar;8(2):131-40. PMID 6857385
- [Background] Walker BF. The prevalence of low back pain: a systematic review of the literature from 1966 to 1998. J Spinal Disord. 2000 Jun;13(3):205-17. doi: 10.1097/00002517-200006000-00003. PMID 10872758